CLINICAL TRIAL: NCT05951647
Title: The Effect of Mouthwashes Containing Pomegranate Peel, German Chamomile or Their Combination in the Treatment of Gingivitis
Brief Title: The Effect of Pomegranate Peel, German Chamomile or Their Combination on Gingivitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0107722
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Gingivitis
Keywords: Pomegranate peel; German chamomile; TNF-α; IL-1β
MeSH Terms: conditions — Gingivitis | interventions — Chamomile extract; Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: Double-blinded, parallel, randomized clinical trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Scaling (Placebo Comparator): 12 patients will be managed by scaling only
  Interventions: Procedure: Scaling
- Scaling and Chlorohexidine mouthwash (Active Comparator): Patients will be managed by scaling and will use 0.12%% chlorohexidine mouthwash in a dose of 15 ml twice daily.
  Interventions: Drug: Scaling and Chlorohexidine mouthwash
- Scaling and Chamomile extract mouthwash (Experimental): Patients will be managed by scaling and will use 5% chamomile extract mouthwash in a dose of 15 ml twice daily.
  Interventions: Drug: Chamomile extract mouthwash
- Scaling and Pomegranate peel extract mouthwash (Experimental): Patients will be managed by scaling and will use 5% pomegranate peel extract mouth wash in a dose of 15 ml twice daily.
  Interventions: Drug: Pomegranate peel extract mouth wash
- Scaling and Chamomile extract mixed with Pomegranate peel extract mouthwash (Experimental): Patients will be managed by scaling and will use a combination of 5% chamomile extract and pomegranate peel extract mouthwash in a dose of 15 ml twice daily.
  Interventions: Drug: Combination of 5% chamomile extract and pomegranate peel extract mouthwash

INTERVENTIONS:
Drug: Chamomile extract mouthwash — 5% chamomile extract mouthwash in a dose of 15 ml twice daily.
  Arms: Scaling and Chamomile extract mouthwash
Drug: Pomegranate peel extract mouth wash — 5% pomegranate peel extract mouth wash in a dose of 15 ml twice daily.
  Arms: Scaling and Pomegranate peel extract mouthwash
Drug: Combination of 5% chamomile extract and pomegranate peel extract mouthwash — Use a combination of 5% chamomile extract and pomegranate peel extract mouthwash in a dose of 15 ml twice daily.
  Arms: Scaling and Chamomile extract mixed with Pomegranate peel extract mouthwash
Procedure: Scaling — Patients will be managed by scaling
  Arms: Scaling
Drug: Scaling and Chlorohexidine mouthwash — scaling and will use 0.12%% chlorohexidine mouthwash in a dose of 15 ml twice daily.
  Arms: Scaling and Chlorohexidine mouthwash

SUMMARY:
The aim of this study is to compare clinically and biochemically the effect of herbal mouthwashes containing German chamomile and pomegranate peel extracts individually and as a mixture to chlorohexidine mouthwash in the treatment of gingivitis. The response will be assessed clinically and by suitable biochemical parameters.

DETAILED DESCRIPTION:
1. Ethical committee approval has been obtained from Ethics committee of Faculty of Medicine and Faculty of Dentistry, Alexandria University
2. All participants should agree to take part in this clinical study and will provide informed consent.
3. Sixty plaque induced gingivitis patients ,will be recruited from Faculty of Dentistry, Alexandria University.
4. The 60 participants will be randomly assigned into 5 groups. Group 1: Patients will be managed by scaling. Group 2: Patients will be managed by scaling and will use 0.12%% chlorohexidine mouthwash in a dose of 15 ml twice daily.

   Group 3: Patients will be managed by scaling and will use 5% chamomile extract mouthwash in a dose of 15 ml twice daily.

   Group 4: Patients will be managed by scaling and will use 5% pomegranate peel extract mouth wash in a dose of 15 ml twice daily.

   Group 5: Patients will be managed by scaling and will use a combination of 5% chamomile extract and pomegranate peel extract mouthwash in a dose of 15 ml twice daily.
5. All patients will be submitted to:

   * Full patient history and clinical examination.
   * Gingival index will be measured
   * Saliva samples will be obtained in order to conduct ELISA for the selected biomarkers.
   * Different mouthwashes will be provided to patients.
6. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
7. Results, conclusion, discussion and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25-50
* Patients with plaque induced gingivitis.

Exclusion Criteria:

* Patients with systemic diseases (diabetes, leukemia, anemia)
* Smokers
* Pregnant females
* Patients receiving orthodontic treatment

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-11 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment for the gingival index (GI) | 15 days
  The gingival index will measured before treatment, 7 days, and 15 days after treatment respectively.

SECONDARY OUTCOMES:
Measurement of TNF-α saliva level | 15 days
  TNF-α saliva level will be measured before treatment, 7 days, and 15 days after treatment respectively.
Measurement of IL1β saliva level | 15 days
  IL1β saliva level will be measured before treatment, 7 days, and 15 days after treatment respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Sh Anwar, PhD, Principal Investigator — Faculty of Pharmacy, Alexandria University; Maha R Taalab, PhD, Principal Investigator — Alexandria University; Doaa A Ghareeb, PhD, Principal Investigator — Faculty of Science, Alexandria University; Noha A Hamdy, PhD, Principal Investigator — Faculty of Pharmacy, Alexandria University; Marwa A Alashwah, PharmD, Principal Investigator — Faculty of Pharmacy, Alexandria University
Locations (1):
- Faculty of Pharmacy, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No